CLINICAL TRIAL: NCT03776032
Title: A Double-Blind, Placebo Controlled, Randomised Study of Novel Erythropoiesis Stimulating Protein (NESP) for the Treatment of Anaemia in Lung Cancer Subjects Receiving Multicycle Platinum-Containing Chemotherapy
Brief Title: A Novel Erythropoiesis Stimulating Protein (NESP; Darbopoetin Alfa) for the Treatment of Anemia in Lung Cancer Patients Receiving Multi-cycle Platinum-Containing Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00980297
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Anemia
Keywords: Lung cancer
MeSH Terms: conditions — Anemia; Lung Neoplasms | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darbepoetin alfa (Experimental): Participants received once a week darbepoetin alfa, administered by subcutaneous injection at a starting dose of 2.25 µg/kg for up to 12 weeks. The dose of darbepoetin alfa may have been adjusted based on hemoglobin levels to a maximum dose of 4.5 µg/kg /week.
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator): Participants received once a week placebo, administered by subcutaneous injection for up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin alfa — Administered by subcutaneous injection once a week
  Other Names: Novel Erythropoiesis Stimulating Protein (NESP); Aranesp
  Arms: Darbepoetin alfa
Drug: Placebo — Placebo matching to darbopoetin alfa administered by subcutaneous injection once a week.
  Arms: Placebo

SUMMARY:
The primary objective of this study was to compare the effectiveness of darbopoetin alfa to placebo in the treatment of anemia in adults with lung cancer receiving multicycle platinum-containing chemotherapy, by assessing the percentage of participants who received red blood cell (RBC) transfusions during weeks 5-12 inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer (either small cell [SCLC] or non-small cell [NSCLC])
* At least 12 additional weeks of platinum containing cyclic chemotherapy planned regardless of cycle length
* Anemia (hemoglobin ≤ 11.0 g/dL) as assessed by a local or central laboratory result within 7 days before study day 1 (the first scheduled day of on-study chemotherapy and the first day of study drug administration)
* Life expectancy of at least 6 months, and an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Anemia predominantly due to the cancer or chemotherapy (i.e.. serum folate ≥ 4.5 nmol/L (≥ 2.0 ng/mL) and vitamin B 12 ≥ 148 pmol/L (≥ 200 pg/mL), no overt hemolysis, and no overt gastrointestinal bleeding or bleeding due to recent surgery)
* Adequate renal function (creatinine ≤ 177gmol/L (≤ 2.0 mg/dL) and adequate hepatic function (bilirubin ≤ 1.5 times central laboratory's upper limit of normal range)
* Available for 4 weeks post administration of the last dose of study drug
* Legal age for informed consent, and written informed consent must be obtained

Exclusion Criteria:

* History of any primary hematological disorder which could cause anemia (e.g., sickle cell anemia)
* Received prior whole pelvis radiation therapy
* Uncontrolled angina, congestive heart failure (New York Heart Association > class II or known ejection fraction < 40%)], or uncontrolled cardiac arrhythmia.
* History of primary or metastatic malignancy involving the central nervous system (CNS). Subjects with a previous history of primary or metastatic malignancy involving the CNS will be eligible for the study providing they have had no clinical signs of nor treatment for CNS disease and no history of seizures within previous 2 years
* Uncontrolled hypertension (i.e., diastolic blood pressure > 100 mm Hg)
* History of seizures. Subjects with a previous history of seizures will be eligible for the study providing they have had no evidence of seizure activity and have been free of anti-seizure medication for the previous 5 years
* Evidence of clinically significant systemic active infection or chronic inflammatory disease (e.g., rheumatoid arthritis)
* Iron deficiency (transferrin saturation < 15% and ferritin < 10 μg/L (< 10 ng/mL))
* Received > 2 RBC transfusions within 4 weeks before randomization or any RBC transfusion within 2 weeks before randomization
* Received erythropoietin therapy within 8 weeks before randomization
* Known positive test for human immunodeficiency virus (HIV) infection
* Receiving, or not yet 30 days past the end of receiving, another investigational agent or device not approved in any indication.
* Pregnant or breast feeding females.
* Not using adequate contraceptive precautions
* Prior treatment with NESP
* Previously randomized in this study
* Known hypersensitivity to mammalian-derived product
* Concerns for subject's compliance with the protocol procedure, including completion of the quality of life surveys (QOLS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 1999-09-14 (Actual); Primary Completion 2000-11-08 (Actual); Study Completion 2002-02-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Red Blood Cell Transfusion During Weeks 5 to 12 | Weeks 5 to 12

SECONDARY OUTCOMES:
Time to First Red Blood Cell Transfusion During Weeks 5 to 12 | Week 5 to week 12
  The number of days from the first day of study week 5 (day 29) to the first administration of a RBC transfusion during the Treatment Phase that occurs on or after day 29.
Percentage of Participants with a Hemoglobin Response by Week 12 | 12 weeks
  Hemoglobin Response was defined as an increase in hemoglobin of ≥ 2.0 g/dL over baseline hemoglobin in the absence of any RBC transfusions during the preceding 28 days.
Time to Hemoglobin Response | 12 weeks
  The number of days from the first administration of study drug to the first occurrence of a hemoglobin response.
Percentage of Participants who Achieved a Sustained Hemoglobin Response by Week 12 | 12 weeks
  Sustained hemoglobin response was defined as in increase in hemoglobin of ≥ 2.0 g/dL over baseline hemoglobin sustained for at least 28 days or until the end of the Treatment Phase. This increase must have occurred in the absence of RBC transfusions during the period of sustained response and the preceding 28 days.
Time to Sustained Hemoglobin Response | 12 weeks
  The number of days from the first administration of study drug to the first occurrence of a sustained hemoglobin response.
Percentage of Participants who Achieved a Hemoglobin Correction by Week 12 | 12 weeks
  Hemoglobin correction was defined as a hemoglobin value of ≥ 12.0 g/dL that occurred in the absence of RBC transfusions during the preceding 28 days.
Percentage of Participants who Achieved a Sustained Hemoglobin Correction by Week 12 | 12 weeks
  Sustained hemoglobin correction was defined as a hemoglobin value of ≥ 12.0 g/dL that was sustained for at least 28 days or until the end of the Treatment Phase. This must have occurred in the absence of RBC transfusions during the period of sustained correction and the preceding 28 days.
Time to Hemoglobin Correction | 12 weeks
  The number of days from the first administration of study drug to the first occurrence of a hemoglobin correction.
Time to Sustained Hemoglobin Correction | 12 weeks
  The number of days from the first administration of study drug to the first occurrence of a sustained hemoglobin correction.
Change from Baseline in Hemoglobin at Week 12 | Baseline and week 12
Percentage of Participants who Received a Red Blood Cell Transfusion During Weeks 1 to 4, 5 to 8, and 9 to 12 | Weeks 1 to 4, 5 to 8, and 9 to 12
Number of Standard Units of RBCs Transfused During Weeks 5 to 12 | Weeks 5 to 12
Number of Days with RBC Transfusions During Weeks 5 to 12 | Weeks 5 to 12
Change from Baseline in the Functional Assessment of Cancer Therapy (FACT)-Anemia Subscales at Week 12 | Baseline and week 12
  The FACT-anemia is a 47-item questionnaire to assess specific quality of life concerns related to anemia and fatigue in cancer patients.
Number of Participants with Adverse Events | 16 weeks